CLINICAL TRIAL: NCT05279157
Title: Implantation of Autologous Mesenchymal Stem Cells of Adipose Origin for the Treatment of Corneal Diseases
Brief Title: Autologous Adipose-Derived Adult Stem Cell Implantation for Corneal Diseases (ADASCs-CT-CD)
Acronym: ADASCs-CT-CD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vissum, Instituto Oftalmológico de Alicante (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EI17-00523; 2018-000523-14 (EudraCT Number)
Record Dates: First submitted 2021-12-17; First posted 2022-03-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Ophthalmological Disorder; Corneal Dystrophy; Treatment; Therapy; Keratoconus
Keywords: Regenerative medicine; Corneal bioengineering; Stem cell therapy; Keratoconus; Adipose-derived adult stem cells (ADASCs); Keratocytes; Corneal confocal microscopy; Advanced corneal therapy
MeSH Terms: conditions — Eye Diseases; Corneal Dystrophies, Hereditary; Keratoconus | interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: In this study, 15 evaluable patients affected by corneal stromal dystrophies of any type (particularly keratoconus) will be included in 3 different groups. Ten patients will be included in the two experimental groups and five in the control group with cell-free treatment (5 patients per group and a total of 3 groups)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients who agree to participate in the study and sign the informed consent will be randomized to enter one of the three groups in a 1: 1: 1 ratio. For this, a randomization scheme will be used that will be unknown to the patient, the center staff, and the promoter staff who intervene directly in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ADASCs Group (Experimental): 5 patients, who will receive adipose tissue mesenchymal stem cells in a single dose as study treatment
  Interventions: Procedure: Implantation; Procedure: Lipoaspiration
- Acellular laminas group (Experimental): 5 patients, who will receive decellularized corneal laminas as treatment medication
  Interventions: Procedure: Implantation
- ADASCs recellularized laminas group (Experimental): 5 patients, who will receive adipose tissue mesenchymal cells combined with decellularized corneal laminas as study treatment in a single intervention
  Interventions: Procedure: Implantation; Procedure: Lipoaspiration

INTERVENTIONS:
Procedure: Implantation — Procedure: Implantation The ophthalmologist will carry out the implantation of the ADASCs cells with or without scaffold in the intrastromal cornea of the patient
  Other Names: corneal implantation
Procedure: Lipoaspiration — Procedure: Lipoaspiration The patient will have a liposuction surgery from which the autologous ADASCs implant in the cornea will be obtained.
  Procedure: Implantation The ophthalmologist will carry out the implantation of the ADASCs with or without scaffold in the intrastromal cornea of the patient
  Other Names: corneal implantation
  Arms: ADASCs Group; ADASCs recellularized laminas group

SUMMARY:
Cellular therapy of the corneal stroma with implantation of mesenchymal stem cells derived from autologous adipose tissue with or without a carrier (scaffold) composed by decellularized human donor corneal stroma is used in patients with corneal diseases such as corneal dystrophies, and keratoconus.

For this purpose, the study planned to assess the enhancement of visual acuity, pachymetric, and aberrometric parameters with implantation of autologous mesenchymal adipose tissue-derived adult stem cells (ADASCs) alone, 120 µm thickness of decellularized or recellularized laminas with ADASCs. Three groups will be included in the study: (1) Implantation of a single dose of ADASCs alone without scaffold. (2) Implantation of decellularized human corneal lamina without ADASCs. (3) Implantation of the recellularized human corneal lamina with ADASCs.

DETAILED DESCRIPTION:
Different types of stem cells have been used in various ways in several research projects to find the optimal procedure to regenerate the human corneal stroma. It included several approaches which can be classified as intrastromal implantation of stem cells (1) alone, (2) together with a biodegradable scaffold, (3) with a non-biodegradable scaffold, or (4) with a decellularized corneal stromal scaffold. The complex structure of the corneal stroma has not been yet replicated, and there are well-known drawbacks to the use of synthetic scaffold-based designs. Recently, several corneal decellularization techniques have been described, which provide an acellular corneal extracellular matrix (ECM). These scaffolds have gained attention in the last few years. The scaffold provides a more natural environment for the growth and differentiation of cells when compared with synthetic scaffolds. In addition, components of the ECM are generally conserved among species and are tolerated well even by xenogeneic recipients. Keratocytes are essential for remodeling the corneal stroma and for normal epithelial physiology. This highlights the importance of transplanting a cellular substitute together with the structural support (acellular ECM) to undertake these critical functions in corneal homeostasis. To the best of the investigators' knowledge, all attempts to repopulate decellularized corneal scaffolds have used corneal cells, but these cells have major drawbacks that preclude their autologous use in clinical practice (damage of the donor tissue, lack of cells, and inefficient cell subcultures), thus the efforts to find an extraocular source of autologous cells. A recent study by the investigators has shown a perfect bio integration of human decellularized corneal stromal laminas (100 µm thickness) with and without h-ADASCs colonization inside the rabbit cornea in vivo, without observing any rejection response despite the graft being xenogeneic. The investigators also demonstrated the differentiation of h-ADASCs into functional keratocytes inside these implants in vivo, which then achieved their proper biofunctionalization. According to the investigator's opinion, the transplant of stem cells together with decellularized corneal ECM would be the best technique to effectively restore the thickness of a diseased human cornea, like in keratoconus. Through this technique, and using extraocular mesenchymal stem cells from patients, it is possible to transform allergenic grafts into functional autologous grafts, theoretically avoiding the risk of rejection.

The process flow is defined as following: (1) the file study: which start by receiving the file of the patient, the file will be forwarded to appointed physicians coordinators for review and submission of medical report, then the medical report will be evaluated within the cell therapy committee and the patient will be asked for clinical examination, and after consultation a reply to the patient with medical decision will follow with an approval or not to be recruited and if yes, a brief report about the procedure will be submitted and explained in details to the patient, a consent form must be signed if the patient agree to be included in the study, (2) the patient admission: which may start by completion of the procedure forms and doing the pre-op evaluation (initial work up defined as a clinical and biological assessment upon C.A.S which may include unaided and best spectacle corrected visual acuity, refraction, slit lamp examination, intraocular pressure, fundoscopy, corneal topography, aberrometry, endothelial cell count (specular microscopy), corneal confocal microscopy, as well as blood tests), all this tests should be effectuated by an specialist and reviewed by an ophthalmologist. Then, a lipoaspiration of the subcutaneous adipose tissue to be performed by a plastic surgeon, sample processing at a cGMP facility for isolation and characterization of the stromal vascular fraction enriched with ADASCs as well as laminas preparing (the quality control assessment will be realized before and after all the steps of the procedure starting from the ADASCs collection to implantation including cell culture, cell quiescence, decellularization of human corneal lamina, recellularization of the laminas with ADASCs, and implantation; the assessment will include cell viability, cell number, cell apoptosis, immunophenotyping, infection, inflammation by analyzing the secreted cytokines from ADASCs, lamina cutting, lamina thickness, immunostaining, confocal microscopy, etc.); (3) the delivery (implantation) which starts by a peribulbar or retrobulbar anesthesia where the patient is placed under operating microscope, followed by a femtosecond laser-assisted mid-stromal lamellar dissection, then the autologous ADASCs or laminas or recellularized laminas will be placed within the pocket, and finally closed by a superior incision closure. The patient will be put under antibiotic/steroids for a defined period and followed by the team at 1 week, 2 weeks, 1 month, 3 months, 6 months.

This protocol of cell therapy will be applied exclusively at VISSUM (Alicante-Spain), Barraquer Ophthalmology Center (Barcelona-Spain), Ramon y Cajal Hospital (Madrid-Spain), Asturias Prince Hospital (Madrid-Spain), and Murcia Hospital (Murcia-Spain), in affiliation with Miguel Hernandez of Elche University (Elche-Spain).

The patient's recruitment will take place: for the lipoaspiration, processing, preparing the cellularized laminas and quality control assessments in VISSUM (Alicante-Spain), Barraquer Ophthalmology Center (Barcelona-Spain), Ramon y Cajal Hospital (Madrid-Spain), and Murcia Hospital (Murcia-Spain). All these steps are managed by VISSUM (Prof. J. ALIO).

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by corneal stromal dystrophies of any type, but particularly keratoconus, showing clear evidence in the ophthalmic examination of the presence and clear expression of the disease and loss of vision as a result of it
* Patients with best-corrected visual acuity less than 0.6
* Absence of chronic or recurrent inflammation in the anterior segment and on the ocular surface.
* Patient suitable to undergo corneal graft surgery under local anesthesia, from a medical point of view.
* Pre-surgical analysis of serum biochemistry and normal hematology.
* Serology for Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), and Hepatitis C (HCV) negative.
* No history of malignancy.
* Normal chest x-ray (Rx).
* Normal urinalysis.
* Normal thyroid exam

Exclusion Criteria:

* Dense and extensive corneal stromal scars with severe involvement of the visual axis and located in the pupillary area, causing a decrease in the best corrected vision to levels of 0.1 or less.
* Distance corrected vision with glasses of 0.7 or greater.
* Extreme corneal thinning with risk of perforation.
* Infection.
* Previous corneal surgeries.
* Moderate or severe dry eye.
* Moderate or severe chronic inflammatory pathology of the ocular surface.
* Previous eye surgery other than cataract.
* Presence of cataract or other severe opacity of the transparent media of the eye that could prevent adequate examination of the fundus.
* Other ophthalmic comorbidity such as glaucoma or uveitis or any that requires the chronic use of topical ocular medication.
* Known and severe coagulation abnormalities.
* Any medical condition that may interfere with causing serious adverse effects during the study.
* Presence of active or inactive corneal neovascularization (CNV) in the eye to be treated
* Any immunodeficiency or systemic autoimmune disease
* Any current or intermittent immunosuppressive therapy or low-dose corticosteroids.
* Renal insufficiency, defined by creatine value> 1.3 mg / dL.
* Serological evidence of hepatitis B, hepatitis C, or HIV infection.
* Pregnant or lactating woman.
* Corrected visual acuity in the eye contralateral to the experimental eye less than 20/40 (0.5)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Improvement in best-corrected distance visual acuity (BCDVA). | at 12 months
  Best-corrected visual acuity (BCDVA) will be studied in Snellen charts by Logmar and the corresponding equivalent in decimal scale.

SECONDARY OUTCOMES:
Increase in corneal thickness. | at 12 months
  Corneal thickness will be evaluated by ultrasonic and optical pachymetry (Scheimpflug corneal topography).
Refractive changes | at 12 months
  Refraction will be studied by refractive subjection performed by a certified good clinical practice technician.
Improvement in anterior corneal surface regularity | at 12 months
  Anterior corneal surface regularity will be evaluated by corneal topography map and analysed by the changes in the Zernike polynomials (third order and fourth order spherical aberration).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L Alio, MD, PhD, Principal Investigator — Universidad Miguel Hernandez, Elche, Spain
Locations (1):
- Jorge L. Alio, Alicante, Spain

REFERENCES:
- [Result] Alio Del Barrio JL, El Zarif M, de Miguel MP, Azaar A, Makdissy N, Harb W, El Achkar I, Arnalich-Montiel F, Alio JL. Cellular Therapy With Human Autologous Adipose-Derived Adult Stem Cells for Advanced Keratoconus. Cornea. 2017 Aug;36(8):952-960. doi: 10.1097/ICO.0000000000001228. PMID 28486314
- [Result] Alio Del Barrio JL, El Zarif M, Azaar A, Makdissy N, Khalil C, Harb W, El Achkar I, Jawad ZA, de Miguel MP, Alio JL. Corneal Stroma Enhancement With Decellularized Stromal Laminas With or Without Stem Cell Recellularization for Advanced Keratoconus. Am J Ophthalmol. 2018 Feb;186:47-58. doi: 10.1016/j.ajo.2017.10.026. Epub 2017 Dec 13. PMID 29103962
- [Result] Alio Del Barrio JL, Arnalich-Montiel F, De Miguel MP, El Zarif M, Alio JL. Corneal stroma regeneration: Preclinical studies. Exp Eye Res. 2021 Jan;202:108314. doi: 10.1016/j.exer.2020.108314. Epub 2020 Oct 24. PMID 33164825
- [Result] Alio JL, Alio Del Barrio JL, El Zarif M, Azaar A, Makdissy N, Khalil C, Harb W, El Achkar I, Jawad ZA, De Miguel MP. Regenerative Surgery of the Corneal Stroma for Advanced Keratoconus: 1-Year Outcomes. Am J Ophthalmol. 2019 Jul;203:53-68. doi: 10.1016/j.ajo.2019.02.009. Epub 2019 Feb 15. PMID 30772348
- [Result] El Zarif M, Alio JL, Alio Del Barrio JL, Abdul Jawad K, Palazon-Bru A, Abdul Jawad Z, De Miguel MP, Makdissy N. Corneal Stromal Regeneration Therapy for Advanced Keratoconus: Long-term Outcomes at 3 Years. Cornea. 2021 Jun 1;40(6):741-754. doi: 10.1097/ICO.0000000000002646. PMID 33591032
- [Result] El Zarif M, A Jawad K, Alio Del Barrio JL, A Jawad Z, Palazon-Bru A, de Miguel MP, Saba P, Makdissy N, Alio JL. Corneal Stroma Cell Density Evolution in Keratoconus Corneas Following the Implantation of Adipose Mesenchymal Stem Cells and Corneal Laminas: An In Vivo Confocal Microscopy Study. Invest Ophthalmol Vis Sci. 2020 Apr 9;61(4):22. doi: 10.1167/iovs.61.4.22. PMID 32301973
- [Result] El Zarif M, Alio Del Barrio JL, Arnalich-Montiel F, De Miguel MP, Makdissy N, Alio JL. Corneal Stroma Regeneration: New Approach for the Treatment of Cornea Disease. Asia Pac J Ophthalmol (Phila). 2020 Dec;9(6):571-579. doi: 10.1097/APO.0000000000000337. PMID 33181549
- [Result] El Zarif M, Alio JL, Alio Del Barrio JL, De Miguel MP, Abdul Jawad K, Makdissy N. Corneal Stromal Regeneration: A Review of Human Clinical Studies in Keratoconus Treatment. Front Med (Lausanne). 2021 Feb 23;8:650724. doi: 10.3389/fmed.2021.650724. eCollection 2021. PMID 33708786
- [Derived] Alio JL. Corneal regeneration: How can we make further progress in corneal surgery with advanced therapies to avoid corneal substitution: ESCRS Binkhorst Medal Lecture 2023. J Cataract Refract Surg. 2025 Nov 1;51(11):1026-1033. doi: 10.1097/j.jcrs.0000000000001745. PMID 41126474